CLINICAL TRIAL: NCT00206323
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Determine the Safety and Efficacy of Topiramate in the Treatment of Tourette Syndrome (CAPSS-176)
Brief Title: A Randomized, Placebo-controlled, Tourette Syndrome Study.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Joseph Jankovic, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-13552
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Topiramate; Pharmaceutical Preparations; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo/sugar pill (Placebo Comparator): Placebo or sugar pill
  Interventions: Drug: placebo/sugar pill
- Topiramate (Active Comparator): Topiramate 25 mg to 200 mg
  Interventions: Drug: Topiramate (drug)

INTERVENTIONS:
Drug: Topiramate (drug) — Topiramate 25 mg titrated to 200 mg
  Other Names: Topamax
  Arms: Topiramate
Drug: placebo/sugar pill — placebo
  Other Names: placebo
  Arms: placebo/sugar pill

SUMMARY:
Previous studies using topiramate in Tourette subjects have shown that with the use of this medication subjects report that their tics get better. The purpose of this study is to study if topiramate improves the symptoms of Tourette syndrome, such as motor tics, or other associated symptoms such as attention or obsessive-compulsive problems.

DETAILED DESCRIPTION:
This study consists of three phases: Screening/Washout Phase, Double-Blind Phase and Taper Phase.

SCREENING/WASHOUT PHASE: Your study doctor or his staff will review with you any medications that you are currently taking and may instruct you, if appropriate, to discontinue taking certain medications. Your study doctor or his staff will explain how long you need to stop taking each drug before you can start the study. Depending on the type of medications you may be taking, the Screening/Washout Visit (Visit 1 of the study) may have to be completed in two visits. The screening/washout phase may take up to 90 days. If you agree to participate, the study doctor or his staff will carry out tests to see if you are eligible for this study. At the Screening/Washout Visit, you will have a medical and psychiatric history review (including medications you have taken for treating Tourette Syndrome) and a physical examination (including sitting blood pressure, pulse, temperature, weight and height). A blood sample will be taken (approximately 2-3 teaspoons) and tested to rule out any abnormalities. You will be asked to give a urine sample that will be tested for drug use and, if you are a female that is capable of having a child, to ensure that you are not pregnant at the time of study entry. The pregnancy test must be negative for you to continue in the study. Additionally, you may not currently be breastfeeding to continue in the study. You will undergo a medical and psychiatric evaluation. You will be asked to answer questions using scales, including one that measures the severity of your symptoms of Tourette Syndrome and one that measures your symptoms, if any, of attention deficit hyperactivity disorder (A-D/HD).

TITRATION/MAINTANENCE PHASE: If you continue to qualify for the study after the Visit 1 tests have been reviewed by the study doctor or his staff and you have completed the washout phase, you will return to your study doctor's office for Visit 2. The length of time between Visit 1 and Visit 2 will depend on the kind of medications you are taking (and may need to stop before entering this study). At Visit 2, you will have your blood pressure, pulse and weight measured. You will be asked to answer questions for the same two scales that you completed at Visit 1. You are asked to return all medication bottles (even if empty, partially used or unused) to each study visit. It is very important for us to be able to check study drug compliance.

You will be asked questions about how you are feeling and if you have started taking any new medications or had changes in other medications you may be taking since your last visit.

If you continue to meet eligibility requirements for the study, you will enter the study. You will be assigned by chance to one of two treatment groups. You may receive either topiramate or placebo (an inactive substance). This makes the assessment of the study drug much fairer. The chances you are receiving the study drug versus placebo are 1 to 1 or equal (50% chance that you will receive topiramate and 50% chance that you will receive placebo).

The study will last approximately 10 weeks. You will begin the study by taking 1 tablet of study medication (topiramate 25 mg or placebo) in the evening. This will be Day 1 of the study. After one week of this phase of the study, your study medication dose will be increased to 2 tablets (topiramate 50 mg or placebo) one tablet in the morning and one in the evening. Your study medication dose may continue to be increased until you have reached the dose level the study doctor determines to be appropriate for you, or, you are taking a maximum dose of 200 mgs per day of study medication (topiramate or placebo). Your study doctor may adjust your study medication dose as necessary. Study medication will be provided in 25 mg tablets of topiramate or placebo. Medication is provided in child-resistant bottles. All bottles should be returned (regardless of whether they are partial, empty or full) at each visit. It is important that you follow your study doctor or his staff's instructions on when and how to take the study medication. You will be expected to visit your study doctor or his staff again on Day 28 (Visit 3), Day 56 (Visit 4) and Day 70 (Visit 5) after beginning treatment. At Visit 5 (Day 70), you will be given instructions about reducing your study medication gradually for the next week.

At each visit, you will have your blood pressure, pulse, temperature and weight measured. You will be asked how you are feeling and if you have started taking any new medications or had changes in other medications you may be taking. At Visits 3 and 5 you will be asked again to answer questions for all of the scales that you completed at Visit 2. At Visits 3, 4 and 5, the study doctor or his staff will complete the scale that assesses the severity of your condition. At Visits 3 and 5, the study doctor or his staff will complete one scale that assesses the severity of your Tourette Syndrome symptoms. At Visits 3, 4 and 5 you will have a urine pregnancy test performed again if you are a female capable of bearing a child. The test must be negative to continue in the study. You will have blood drawn again (approximately one teaspoon) at Visits 3 and 5 to make sure that your liver is functioning properly and that your electrolytes (blood chemistry measurements) are also within normal range. At Visit 5 you will have another physical examination.

You will be called weekly between Visits 2 and 3 (Days 7, 14 and Day 21 of the study) and Visits 3 and 4 (Days 35 and 42 of the study) on the telephone by one of the people working on this study. During these phone calls you will be asked how you are feeling, if you have had any changes in medications you are taking and how you are doing with the study medication.

TAPER PHASE: You will visit the study doctor or his staff again on Day 77 (Visit 6) after you have completely stopped taking the study medication. You must keep all medication packaging and any unused medication, and bring it back to the study doctor or his staff at each visit. At this visit, you will have your blood pressure and pulse taken and your weight measured. You will be asked again to answer questions for the scale that measures the severity of your symptoms of Tourette Syndrome. If you are a female capable of bearing a child, a urine pregnancy test will be performed. You will be asked how you are feeling and if you have started taking any new medications or had changes in other medications you may be taking.

Joseph Jankovic, Joohi Jimenez-Shahed and Lawrence Brown J. Neurol. Neurosurg. Psychiatry published online 1 Sep 2009; doi:10.1136/jnnp.2009.185348

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of Tourette Syndrome for at least 3 months.
* Subjects must have a minimum Tic rating scale of > or equal to 19 (current symptoms excluding impairment) at Visit 1 (Day -10 through Day -7) and Visit 2 (Day ).
* Subjects must have a rating scale severity score of > or equal to 4 (moderately ill) at Visit 1 (Day -10 through Day -7) and Visit 2 (Day 1).
* Subjects must be between 7 and 65 years of age, inclusive.
* Subjects must be >25 kg (55 lbs).
* Subjects must be able to take oral medication in tablet form without crushing or otherwise altering the tablet, adhere to medication regimens and be willing to return for regular visits.
* Subjects must have observed the designated washout periods for prohibited medications outlined under the Concomitant Therapy section of this protocol.
* Subjects must have a negative urine drug screening at Visit 1 (Day -7).
* Subjects must be in generally good health as confirmed by medical history, baseline psychiatric history and physical examination, including vital signs.
* Subjects must: a) be premenarchal, postmenopausal for at least one year, or b) have had a hysterectomy or tubal ligation or otherwise be incapable of pregnancy, or c) have practiced one of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, spousal/partner sterility or d) be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence. If (c) or (d), subjects must have a negative urine pregnancy test up to one week prior to Visit 2 (Day 1).
* Subjects, or their parents/guardians, must be able to read and comprehend written instructions and willing to complete all scales and inventories required by this protocol.

Exclusion Criteria:

* Subjects who have a diagnosis of substance dependence or abuse (with the exception of nicotine or caffeine dependence) within the past 3 months.
* Subjects with a significant and unstable major psychiatric disorder requiring treatment.
* Subjects with mental retardation.
* Subjects with progressive or degenerative neurological disorders or a structural disorder of the brain from birth, trauma or past infection.
* Subjects taking more than one agent for the treatment of tics, more than one agent for the treatment of comorbid symptoms or more than one agent for the treatment of ADHD and/or the dose of the current treatment has not been stable for a minimum of 6 weeks.
* Subjects who are pregnant or lactating.
* Subjects with prior non-response to topiramate for the treatment of Tourette Syndrome following an adequate trial.
* Subjects with a history of nephrolithiasis.
* Subjects with an estimated creatinine clearance of <60 mL/min.
* Subjects who have Liver function levels greater than 2 times the upper limit of the normal range at Visit 1.
* Subjects who have active liver disease.
* Subjects who have previously been treated with topiramate and discontinued treatment due to an adverse event or subjects with a known hypersensitivity to topiramate.
* Subjects known to have clinically significant medical conditions, including, but not limited to: a) any unstable disease or condition, including cardiovascular, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease that could compromise the function of those body systems that could result in altered absorption, excess accumulation or impaired metabolism or excretion of topiramate or interfere with their participation in the study; b) malignancy or history of malignancy (excluding basal cell carcinoma) within the past 5 years; and c) subjects with a history of attempted suicide or suicidal tendencies or judged clinically to be at serious suicidal risk

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jankovic, MD, Principal Investigator — Baylor College of Medicine

REFERENCES:
- [Background] Jankovic J, Jimenez-Shahed J, Brown LW. A randomised, double-blind, placebo-controlled study of topiramate in the treatment of Tourette syndrome. J Neurol Neurosurg Psychiatry. 2010 Jan;81(1):70-3. doi: 10.1136/jnnp.2009.185348. Epub 2009 Sep 1. PMID 19726418

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: Topiramate versus placebo
  Topiramate (drug): Topiramate 25 mg titrated to 200 mg
Period: Overall Study
Arm/Group | Placebo/Sugar Pill | Topiramate
Started | 14 | 15
Completed | 8 | 12
Not Completed | 6 | 3
Not completed — Lack of Efficacy | 4 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Sugar Pill | Topiramate | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 15 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age 7-65 with DSM-IV criteria for Tourette Syndrome to be enrolled in study.
  years | 14.1 (8.35) | 18.8 (10.93) | 16.5 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Tic Score at Day 70
Description: A component of the Yale Global Tic Severity Scale (YGTSS), the change from baseline in Total Tic Score (TTS) at visit 5 (day 70) is the pre-defined primary endpoint.
  The Total Tic Score (TTS) is a summation of the Total Motor Tic and Total Phonic Tic Scores. The Overall Impairment Rating is rated on a 50-point scale anchored by 0 (No impairment) and 50 (Severe impairment).
Time Frame: baseline and Day 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo/Sugar Pill | Topiramate
Number analyzed (Participants) | 13 | 14
units on a scale | -5.0 (9.88) | -14.29 (10.47)
Statistical Analysis 1: Comparison: Placebo/Sugar Pill vs Topiramate; Primary variable change of TTS/YGTSS at the BSL to Day 70. Changes of YGTSS compared using analysis of covariance with score at day 1 as a covariate. Groups compared for incidence of AE's and of AESI based on Fisher's Exact Test. All tests were two-sided at the 5% level of significance. The Total Tic Score is a summation of the Total Motor Tic and Total Phonic Tic Scores. The Overall Impairment Rating is rated on a 50-point scale anchored by 0 (No impairment) and 50 (Severe impairment); Test type: Superiority or Other; p = 0.0259, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo/Sugar Pill | Topiramate
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 8/14 | 11/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Sugar Pill (N=14) | Topiramate (N=15)
headache (General disorders) | 3 (3) | 3 (3)
diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
drowsiness (General disorders) | 2 (2) | 2 (2)
cognitive slowing (General disorders) | 0 (0) | 1 (1)
kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No